Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625 Reparto Tel 02/55033789 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a> U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio Tel. 02 55032503 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

## STUDY PROTOCOL

The Italian REgistry of pulmonary Non-tuberculous mycobactEria – IRENE

Version #: 2.0

Date: June 21<sup>st</sup>, 2017



/02/50320625

Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare

U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a>

U.O.S Fibrosi Cistica Sez. Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

**Study Sponsor:** 

UO di Broncopneumologia, Dipartimento delle Units multispecialistiche e dei trapianti / Area

Cardio-Polmonare, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano

**Principal Investigator:** 

• Prof. Stefano Aliberti, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti,

Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units

multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda

Ospedale Maggiore Policlinico, Milano; E-mail: stefano.aliberti@unimi.it.

**Executive committee:** 

Prof. Stefano Aliberti, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti,

Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units

multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda

Ospedale Maggiore Policlinico, Milano; E-mail: stefano.aliberti@unimi.it.

• Prof. Francesco Blasi, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti,

Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units

/02/50320625

Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <u>broncopneumologia@policlinico.mi.it</u>

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda

Ospedale Maggiore Policlinico, Milano; E-mail: francesco.blasi@unimi.it.

• Dr. Luigi Ruffo Codecasa, Centro regionale di riferimento per TB, Istituto Villa Marelli, ASST

Grande Ospedale Metropolitano Niguarda, Milano; E-mail:

luigiruffo.codecasa@ospedaleniguarda.it

Prof. Andrea Gori, Scuola di Medicina e Chirurgia, Università degli Studi di Milano Bicocca,

UO Malattie Infettive, ASST di Monza, Ospedale San Gerardo, Monza; E-Mail:

andrea.gori@unimib.it

**Scientific Committee** 

1. Prof. Stefano Aliberti, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti,

Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units

multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda

Ospedale Maggiore Policlinico, Milano

2. Prof. Francesco Blasi, Dipartimento di Fisiopatologia Medico-Chirurgica e dei Trapianti,

Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units

multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda

Ospedale Maggiore Policlinico, Milano

Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625 Reparto Tel 02/55033789 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a> U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio Tel. 02 55032503 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

- 3. Dr. Luigi Ruffo Codecasa, Centro regionale di riferimento per TB, Istituto Villa Marelli, ASST Grande Ospedale Metropolitano Niguarda, Milano
- Prof. Andrea Gori, Scuola di Medicina e Chirurgia, Università degli Studi di Milano Bicocca,
  UO Malattie Infettive, ASST di Monza, Ospedale San Gerardo, Monza
- 5. Prof. Giovanni Sotgiu, Clinical Epidemiology and Medical Statistics Unit, Department of Biomedical Sciences, Università degli Studi di Sassari, Sassari, Italia
- 6. Dr Stefano Nardini, UO di Pneumotisiologia, Ospedale di Vittorio Veneto, Treviso, Italia
- 7. Dr Mehdi Mirsaeidi, Division of Pulmonary and Critical Care, University of Miami, 1600 NW, Miami, FL 33136, USA; Miami VA Medical Center, 1201 N.W. 16th St., Miami, FL 33125, USA.
- 8. Dr Enrico Tortoli, Emerging Bacterial Pathogens Unit, IRCCS Ospedale San Raffaele, Milano, Italia
- 9. Dr Giorgio Besozzi, Stop TB Italia, Milano, Italia
- 10. Dr Alberto Matteelli, Clinic of Infectious and Tropical Diseases, University of Brescia and Brescia Spedali Civili General Hospital, WHO Collaborating Centre for TB/HIV and TB Elimination, Brescia, Italia
- 11. Dr Antonio Di Biagio, IRCCS-AOU-San Martino-IST, Infectious Disease Clinic, Genova, Italia
- 12. Dr Andrea Calcagno, Università degli Studi di Torino

Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625 Reparto Tel 02/55033789 Fax 02/55034150 Mail: <a href="mailto:broncopneumologia@policlinico.mi.it">broncopneumologia@policlinico.mi.it</a> U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio Tel. 02 55032503 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

- 13. Dr Girardi Spallanzani, UOC Epidemiologia Clinica Dipartimento di Epidemiologia e Ricerca Preclinica, Clinical Epidemiology Unit Department of Epidemiology and Preclinical Research Istituto Nazionale Malattie Infettive "L. Spallanzani" IRCCS Via Portuense 292, 00149 Roma
- 14. Dr Giuliana Previdi, rappresentate pazienti
- 15. Dr Baroukh Maurice Assael, Università degli Studi di Milano, UO di Broncopneumologia, Dipartimento delle Units multispecialistiche e dei trapianti / Area Cardio-Polmonare, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano

/02/50320625

Dipartimento delle Units multispecialistiche e dei Trapianti – Area Cardiopolmonare U.O.C. Broncopneumologia - Direttore: Prof Francesco Blasi

Direzione Tel. 02 55033781-2/02 50320627-3 Fax 02/50320625

Reparto Tel 02/55033789 Fax 02/55034150 Mail: <u>broncopneumologia@policlinico.mi.it</u>

U.O.S Fibrosi Cistica Sez . Adulti – Responsabile: Dr.ssa Giovanna Pizzamiglio

Tel. 02 55032503 Fax 02/55034150 Mail: broncopneumologia@policlinico.mi.it

**STATISTICAL ANALYSIS** 

All statistical analyses will be performed with SPSS (version 17.0) for Mac. A descriptive statistical

analysis at baseline will be performed and results will be reported as mean (± SD) for scale

variables and as counts (%) for nominal variables. The proportion of patients with NTM-PD who

will be treated and managed according to the recommendations published by the latest

international guidelines will be reported: the numerator will be the number of patients with NTM-

PD treated according to those recommendations, while the denominator will be the total number

of patients with NTM-PD[1].

**REFERENCES** 

1. Haworth CS, Banks J, Capstick T, Fisher AJ, Gorsuch T, Laurenson IF, Leitch A, Loebinger MR, Milburn HJ, Nightingale M, Ormerod P, Shingadia D, Smith D, Whitehead N, Wilson R, Floto RA. British Thoracic Society guidelines for the management of non-tuberculous

mycobacterial pulmonary disease (NTM-PD). Thorax. 2017 Nov;72(Suppl 2):ii1-ii64.